CLINICAL TRIAL: NCT05810545
Title: Drinking Water PFAS, Pregnancy Outcome and Maternal Morbidity
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council for Environment, Agricultural Sciences and Spatial Planning (FORMAS) (Other Government); The Swedish Research Council (Other Government); Statistics Sweden (Unknown); National Board of Health and Welfare, Sweden (Other Government); Swedish University of Agricultural Sciences (Other); Swedish Food Agency (Unknown)
Responsible Party: Principal Investigator, Agneta Åkesson, Professor, Karolinska Institutet
Other Study IDs: EXP-21-CV8301; 2022-00980 (Other Grant/Funding Number: Swedish Research Council)
Record Dates: First submitted 2023-03-31; First posted 2023-04-12 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Birth Weight; Small for Gestational Age at Delivery; Large for Gestational Age at Delivery (Macrosomia); Diabetes, Gestational; Hypertension in Pregnancy; Preeclampsia; Congenital Malformation
MeSH Terms: conditions — Birth Weight; Diabetes, Gestational; Hypertension, Pregnancy-Induced; Pre-Eclampsia; Congenital Abnormalities | interventions — Fluorocarbons

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Per- and polyfluoroalkyl substances (PFAS) — Assess the association between exposure to per- and polyfluoroalkyl substances (PFAS) via drinking water in pregnancy and birth outcomes (i.e. growth retardation, premature birth, and congenital developmental defects) and maternal morbidity (gestational hypertension, diabetes and preeclampsia) in a prospective population-wide register based cohort.

SUMMARY:
The aim of the project is to assess the association between exposure to per- and polyfluoroalkyl substances (PFAS) via drinking water in pregnancy and birth outcomes (i.e. growth retardation, premature birth, and congenital developmental defects) and maternal morbidity (gestational hypertension, diabetes and preeclampsia) in a prospective population-wide register study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women residing in Swedish localities with a population exceeding 10,000 inhabitants and giving birth during 2012-2018

Exclusion Criteria:

* Lack of data of PFAS levels in municipal drinking water (entire localities excluded)
* Mothers not living in the study area consistently between first trimester and four years prior to birth

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women residing in Swedish localities with a population exceeding 10,000 inhabitants and giving birth during 2012-2018, where PFAS exposure data is available.
Sampling Method: Probability Sample
Enrollment: 256659 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Birth outcome - birthweight | at birth
  grams as measured at birth
Birth outcome - Small for gestational age (SGA) | at birth
  <-2 standard deviations (SD) from the average weight at the gestational age and sex at partus (Marsal et al. 1996. Acta Paediatr 85(7): 843-848)
Birth outcome - Large for gestational age (LGA) | at birth
  >2 standard deviations (SD) from the average weight at the gestational age and sex at partus (Marsal et al. 1996. Acta Paediatr 85(7): 843-848)
Birth outcome - major congenital malformations | at birth
  ICD10- codes: Q00-Q99 within the first 28 days postpartum, categorized as major congenital malformations according to European Surveillance of Congenital Anomalies (EUROCAT 2014)
Maternal health - Gestational hypertension/preeclampsia | during gestation
  ICD10-codes: O13-O14. Diagnosis at maternal or primary care
Maternal health - Gestational diabetes mellus | during gestation
  ICD10-codes: O24 (excluding pregestational diabetes). Diagnosis at maternal or primary care

IPD SHARING:
Plan to Share IPD: No
IPD is available from registers at Statistics Sweden and National Board of Health and Welfare in Sweden.